CLINICAL TRIAL: NCT00488683
Title: A Phase II, Single Center, Open-label, Randomized Study to Investigate Meningococcal Serogroup A, C, W-135 and Y Saccharide Specific B Cell Response to a Primary and a Booster Course of the Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Infants
Brief Title: B Cell Response to a Primary and a Booster Course of the Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P16; 2006-003476-35
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal disease; Prevention; Vaccination
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY-CRM vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Tetanus Toxoid; Poliovirus Vaccine, Inactivated; Heptavalent Pneumococcal Conjugate Vaccine; Rubella Vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MenACWY-CRM and Routine Vaccines (Group 1) (Experimental): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 13 months), and 1 dose each of MMR and Hib (booster) at 13 months.
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-Hib-IPV; Biological: PCV; Biological: MMR; Biological: Hib
- MenACWY-CRM and Routine Vaccines (Group 2) (Experimental): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 12 months), and 1 dose each of MMR and Hib (booster) at 13 months.
  This group had an additional blood draw at the time of enrollment.
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-Hib-IPV; Biological: PCV; Biological: MMR; Biological: Hib
- MenACWY-CRM and Routine Vaccines (Group 3) (Experimental): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 12 months), and 1 dose each of MMR and Hib (booster) at 13 months of age.
  This group had an additional blood draw at 6-7 days after third dose of MenACWY-CRM.
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-Hib-IPV; Biological: PCV; Biological: MMR; Biological: Hib

INTERVENTIONS:
Biological: MenACWY-CRM — One dose (0.5 mL) of MenACWY conjugate vaccine supplied as an extemporaneous mixing just before injection of the lyophilized component (MenA) reconstituted with the liquid component (MenCWY) was administered at 2-, 4-, and 12-months as IM injections in the anterolateral area of the right thigh.
Biological: DTaP-Hib-IPV — IM injections of 3 doses of 0.5 mL each of DTaP-Hib-IPV supplied in prefilled vial were administered at 2-, 3-, and 4-months in the anterolateral area of the left thigh.
  Other Names: Combined diphtheria, tetanus toxoid, acellular pertussis, Haemophilus influenzae type B and inactivated polio vaccine; Pediacel
Biological: PCV — IM injections of 3 doses of 0.5 mL each of PCV supplied in pre-filled syringe were administered at 2-, 4-, and 12-months (Groups 2 and 3) or 13-months (Group 1) in the anterolateral area of the left thigh.
  Other Names: Heptavalent Streptoccus pneumonia; Prevnar
Biological: MMR — IM injection of one dose of 0.5 mL of MMR obtained by extemporaneous mixing just before injection of powder and the solvent for solution was administered at 13 months in the anterolateral area of the left thigh.
  Other Names: Measles, mumps, and rubella vaccine; Priorix
Biological: Hib — IM injection of one dose 0.5 mL of Hib supplied in pre-filled syringe was administered at 13 months in the anterolateral area of the right thigh.
  Other Names: Vaxem Hib

SUMMARY:
This study is aimed to assess whether the frequency of meningococcal serogroup A, C, W-135 and Y specific memory B Cells, measured 1 month after a primary vaccination series of Novartis MenACWY vaccine, predicts the specific serum bactericidal activity using human complement (hSBA) of (respectively) serogroup A, C, W-135 and Y at 12 months of age

ELIGIBILITY:
Inclusion Criteria:

Subjects who were eligible to be enrolled in the study:

* healthy infants aged 2 months (56 - 83 days old, inclusive);
* available for the visits scheduled in the study;
* mother available for blood draw at Visit 1;
* good health as determined by the clinical judgement of the investigator;
* whose parents gave written informed consent for the infant to be enrolled in the study. The infant's parents must have been willing for the infant to receive the full primary immunization course.

Exclusion Criteria:

Subjects who were not eligible for the study were those:

* whose parents had not given or were unwilling or unable to give written informed consent to their child's participation in the study
* with known hypersensitivity to any vaccines contained within the routine immunization schedule
* with unacceptable concurrent illnesses or conditions - e.g.:

  1. a severe acute or chronic illness; with any present or suspected serious disease such as metabolic, cardiac or autoimmune disease or insulin dependent diabetes or with any other serious disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
  2. a genetic anomaly, e.g. Down's syndrome;
  3. any immunodeficiency, including use of systemic corticosteroids;
  4. born at less than 36 weeks gestation;
  5. weighing less than 2.5 kg at birth;
  6. previous clinical or bacteriological diagnosis of meningitis, or with a history of household contact or intimate exposure to an individual with culture proven Neisseria meningitidis disease;
  7. known bleeding diathesis, or any condition associated with a prolonged bleeding time;
* who have received any prohibited prior or concomitant medications - e.g.:

  1. any immunizations within the 30 days prior to enrollment, with the exception of BCG or hepatitis B;
  2. immunoglobulin;
  3. any blood products;
* participating in any other clinical trial either currently or in the previous month;
* unable to adhere to the protocol, including plans to move from the area;
* Other:

Had any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 56 Days to 83 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Headington, Oxford, United Kingdom

REFERENCES:
- [Result] Blanchard-Rohner G, Snape MD, Kelly DF, O'Connor D, John T, Clutterbuck EA, Ohene-Kena B, Klinger CL, Odrljin T, Pollard AJ. The B-cell response to a primary and booster course of MenACWY-CRM(1)(9)(7) vaccine administered at 2, 4 and 12 months of age. Vaccine. 2013 May 7;31(20):2441-8. doi: 10.1016/j.vaccine.2013.03.036. Epub 2013 Apr 6. PMID 23566945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one study center in the UK.
Pre-assignment Details: All enrolled subjects were included in the trial.
Period: Overall Study
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Started | 108 | 54 | 54
Completed | 96 | 48 | 52
Not Completed | 12 | 6 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Lost to Follow-up | 5 | 3 | 0
Not completed — Protocol Violation | 5 | 1 | 0
Not completed — Unable to Classify | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3) | Total
Number analyzed (Participants) | 108 | 54 | 54 | 216
Age, Continuous [Mean (Standard Deviation); unit: Days] | 60.5 (3.7) | 59.8 (3.6) | 59.8 (3.6) | 60.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 28 | 25 | 101
  Male | 60 | 26 | 29 | 115
Race/Ethnicity, Customized [Number; unit: Subjects]
  Caucasians | 95 | 47 | 51 | 193
  Black | 2 | 2 | 0 | 4
  Asian | 1 | 1 | 0 | 2
  Others | 10 | 4 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Summary of Memory B Cells Per 2 x 105 LOC by Serogroup A, C, W-135 and Y
Description: The memory B cell response at one month after primary vaccinations (5 months of age) was defined as the mean number of meningococcal serogroup A, C, W-135 and Y specific memory B cells, measured in vitro by ELISpot assay per 2x100000 lymphocytes obtained from culture (LOC) of peripheral blood mononuclear cells (PBMC) circulating in blood incubated for 5.5 days in the presence of polyclonal B cell activators.
  Serogroup A, C, W-135 and Y geometric mean titers (GMTs) were measured by serum bactericidal assay using human complement (hSBA) at 12 months of age (before third dose).
  Correlation and linear regression coefficients were determined between memory B cells at 1 month after primary vaccinations with MenACWY-CRM (5 months of age) and hSBA titers at 12 months of age (before third dose) for the serogroups A, C, W-135 and Y.
Time Frame: 1 month after primary vaccination and immediately before third dose at 12 months of age
Population: Analysis was performed on per-protocol (PP) dataset of primary vaccination, i.e. subjects who received all the relevant doses of vaccine correctly; provided evaluable blood samples at the relevant time points; and had no major protocol violation as defined prior to analysis.
Measure: Mean (Standard Deviation); unit: B cells per 2x100000 lymphocytes
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 88 | 34 | 50
B cells per 2x100000 lymphocytes
  Serogroup A (N=50,25,30) | 2.10 (2.03) | 1.80 (1.27) | 1.72 (1.89)
  Serogroup C (N=71,31,43) | 2.57 (2.73) | 1.71 (1.12) | 2.43 (2.32)
  Serogroup W-135 (N=62,26,40) | 2.39 (4.69) | 1.50 (0.721) | 1.57 (1.47)
  Serogroup Y (N=54,25,30) | 2.91 (8.36) | 1.43 (0.71) | 1.78 (1.67)
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.69, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = -0.06
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.30, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.14
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p < 0.0001, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.81
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup Y; Test type: Superiority or Other; p = 0.001, Parametric correlation — Values from Groups I, II and III were combined for this analysis; Pearson correlation coefficient = 0.67
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.61, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = -0.08
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.02, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.31
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p = 0.002, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.45
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup Y; Test type: Superiority or Other; p = 0.08, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.40
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.004
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.02
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.66
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and hSBA titers at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.45

2. Secondary Outcome: Memory B Cells by Serogroup A, C, W-135 and Y
Description: Memory B cell response at 1 month after primary vaccination and immediately before third dose at 12 months of age was measured as mean number of meningococcal serogroup specific memory B cells by ELISpot assay per 2x100000 LOC.
  The meningococcal serogroup A, C, W-135 and Y specific IgG concentrations immediately before third dose at 12 months of age were measured by ELISA.
Time Frame: 1 month after primary vaccination and immediately before third dose
Population: Analysis was performed on PP dataset of persistence population.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 79 | 37 | 39
Value | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.70, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = -0.07
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.37, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = -0.13
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p < 0.0001, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.66
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup Y; Test type: Superiority or Other; p < 0.0001, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.90
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.94, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.01
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.70, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = -0.05
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p = 0.04, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.30
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup Y; Test type: Superiority or Other; p = 0.004, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.46
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.005
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.02
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.43
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and memory B cells at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.82
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.68, Parametric correlation — Values from Group 1, 2 and 2 were combined for this analysis; Pearson correlation coefficient = 0.05
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.46, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.08
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p = 0.08, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.20
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup Y; Test type: Superiority or Other; p < 0.001, Parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Pearson correlation coefficient = 0.45
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup A; Test type: Superiority or Other; p = 0.75, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = -0.04
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup C; Test type: Superiority or Other; p = 0.27, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.11
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup W-135; Test type: Superiority or Other; p = 0.07, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.20
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup Y; Test type: Superiority or Other; p = 0.06, Non-parametric correlation — Values from Group 1, 2 and 3 were combined for this analysis; Spearman correlation coefficient = 0.23
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.0029
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.0059
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.04
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccinations and serogroup specific IgG concentration at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear — Values from Group 1, 2 and 3 were combined for this analysis; R-square = 0.21

3. Secondary Outcome: Memory B Cells Per 2x100000 by Serogroup A,C, W-135 and Y at One Month After Primary MenACWY-CRM Vaccination and Third MenACWY-CRM Vaccination
Description: Memory B cell response at 1 month after MenACWY-CRM primary and booster vaccinations was measured as mean number of meningococcal serogroup specific memory B cells by ELISpot assay per 2x100000 LOC.
  hSBA GMTs for the serogroup A, C, W-135 and Y were measured one month after the third MenACWY-CRM vaccination.
  The meningococcal serogroup A, C, W-135 and Y specific IgG concentrations one month after third MenACWY-CRM vaccination were measured by ELISA.
Time Frame: 1 month after primary vaccination and 1 month after third vaccination
Population: Values from Group 1 were analyzed separately. Values from Groups 2 and 3 were combined for the analysis. Groups 2 and 3 received PCV at 12 months while Group 1 received PCV at 13 months.
  Analysis was performed on PP booster population.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
Value | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.46, Parametric correlation; Pearson correlation coefficient = -0.26
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.59, Parametric correlation; Pearson correlation coefficient = -0.14 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.98, Parametric correlation; Pearson correlation coefficient = 0.006
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.20, Parametric correlation; Pearson correlation coefficient = 0.24 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.08, Parametric correlation; Pearson correlation coefficient = 0.43
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.68, Parametric correlation; Pearson correlation coefficient = -0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.006, Parametric correlation; Pearson correlation coefficient = 0.77
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.48, Parametric correlation; Pearson correlation coefficient = 0.16 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.46, Non-parametric correlation; Spearman correlation coefficient = -0.26
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.40, Non-parametric correlation; Spearman correlation coefficient = -0.21 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.60, Non-parametric correlation; Spearman correlation coefficient = 0.12
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; p = 0.03, Non-parametric correlation; Spearman correlation coefficient = 0.40 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.001, Non-parametric correlation; Spearman correlation coefficient = 0.72
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 1.00, Non-parametric correlation; Spearman correlation coefficient = 0.000 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.24, Non-parametric correlation; Spearman correlation coefficient = 0.39
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 15]; Test type: Superiority or Other; p = 0.34, Non-parametric correlation; Spearman correlation coefficient = 0.22 — Values from Group 2 and 3 were combined for the analysis
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.07
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.000
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 19]; Test type: Superiority or Other; Regression, Linear; R-square = 0.06 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.19
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; Regression, Linear; R-square = 0.007 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.59
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 23]; Test type: Superiority or Other; Regression, Linear; R-square = 0.03 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 25: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.0002, Parametric correlation; Pearson correlation coefficient = 0.77
Statistical Analysis 26: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.90, Parametric correlation; Pearson correlation coefficient = 0.03 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 27: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.02, Parametric correlation; Pearson correlation coefficient = 0.47
Statistical Analysis 28: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 27]; Test type: Superiority or Other; p = 0.12, Parametric correlation; Pearson correlation coefficient = 0.29 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 29: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.22, Parametric correlation; Pearson correlation coefficient = 0.31
Statistical Analysis 30: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; p < 0.0001, Parametric correlation; Pearson correlation coefficient = 0.81 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 31: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.82, Parametric correlation; Pearson correlation coefficient = 0.15
Statistical Analysis 32: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 31]; Test type: Superiority or Other; p = 0.66, Parametric correlation; Pearson correlation coefficient = -0.15 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 33: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.03, Non-parametric correlation; Spearman correlation coefficient = 0.51
Statistical Analysis 34: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; p = 0.53, Non-parametric correlation; Spearman correlation coefficient = 0.14 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 35: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.35, Non-parametric correlation; Spearman correlation coefficient = 0.20
Statistical Analysis 36: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 35]; Test type: Superiority or Other; p = 0.09, Non-parametric correlation; Spearman correlation coefficient = 0.47 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 37: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.04, Non-parametric correlation; Spearman correlation coefficient = 0.51
Statistical Analysis 38: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; p = 0.10, Non-parametric correlation; Spearman correlation coefficient = 0.35 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 39: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.56, Non-parametric correlation; Spearman correlation coefficient = 0.35
Statistical Analysis 40: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 39]; Test type: Superiority or Other; p = 0.84, Non-parametric correlation; Spearman correlation coefficient = -0.07 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 41: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.59
Statistical Analysis 42: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; Regression, Linear; R-square = 0.001 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 43: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.22
Statistical Analysis 44: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 43]; Test type: Superiority or Other; Regression, Linear; R-square = 0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 45: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.10
Statistical Analysis 46: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 45]; Test type: Superiority or Other; Regression, Linear; R-square = 0.66 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 47: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.02
Statistical Analysis 48: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 47]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 49: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.08, Parametric correlation; Pearson correlation coefficient = 0.29
Statistical Analysis 50: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 49]; Test type: Superiority or Other; p = 0.74, Parametric correlation; Pearson correlation coefficient = 0.05 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 51: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.94, Parametric correlation; Pearson correlation coefficient = -0.01
Statistical Analysis 52: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 51]; Test type: Superiority or Other; p = 0.51, Parametric correlation; Pearson correlation coefficient = -0.09 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 53: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.12, Parametric correlation; Pearson correlation coefficient = 0.27
Statistical Analysis 54: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 53]; Test type: Superiority or Other; p = 0.09, Parametric correlation; Pearson correlation coefficient = 0.25 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 55: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.81, Parametric correlation; Pearson correlation coefficient = -0.05
Statistical Analysis 56: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 55]; Test type: Superiority or Other; p = 0.07, Parametric correlation; Pearson correlation coefficient = 0.28 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 57: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.02, Non-parametric correlation; Spearman correlation coefficient = 0.36
Statistical Analysis 58: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 57]; Test type: Superiority or Other; p = 0.59, Non-parametric correlation; Spearman correlation coefficient = 0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 59: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.51, Non-parametric correlation; Spearman correlation coefficient = -0.1
Statistical Analysis 60: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 59]; Test type: Superiority or Other; p = 0.9, Non-parametric correlation; Spearman correlation coefficient = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 61: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.02, Non-parametric correlation; Spearman correlation coefficient = 0.39
Statistical Analysis 62: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 61]; Test type: Superiority or Other; p = 0.20, Non-parametric correlation; Spearman correlation coefficient = 0.19 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 63: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.34, Non-parametric correlation; Spearman correlation coefficient = 0.18
Statistical Analysis 64: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 63]; Test type: Superiority or Other; p = 0.04, Non-parametric correlation; Spearman correlation coefficient = 0.33 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 65: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.08
Statistical Analysis 66: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 65]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0027 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 67: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.0002
Statistical Analysis 68: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 67]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0077 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 69: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.07
Statistical Analysis 70: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 69]; Test type: Superiority or Other; Regression, Linear; R-square = 0.06 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 71: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.0023
Statistical Analysis 72: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 3, analysis 71]; Test type: Superiority or Other; Regression, Linear; R-square = 0.08 — Values from Group 2 and 3 were combined for this analysis

4. Secondary Outcome: Memory B Cells 1 Month After Primary Vaccination and Rise From Pre-third Dose to 1 Month After Third Dose of MenACWY-CRM Vaccination
Description: Memory B cell response at 1 month after MenACWY-CRM primary and third (booster) vaccination was measured as mean number of meningococcal serogroup specific memory B cells by ELISpot assay per 2x100000 LOC.
  The serogroup A, C, W-135 and Y specific IgG concentrations at 1 month after MenACWY-CRM booster were measured by ELISA.
  hSBA GMTs were measured by hSBA assay one month after MenACWY-CRM booster vaccination.
  The rise in serogroup specific IgG, memory B cells and hSBA was calculated by pre/post third dose geometric mean ratios, calculated by the difference in the log10 of the concentrations/titers measured at 13 months to the log10 of the concentrations at 12 months: i.e. rise = log10(x) at 13 months minus log10(x)at 12 months where x is the serogroup specific IgG or memory B cell concentrations or SBA titers.
Time Frame: 1 month after primary and pre-third and 1 month after third vaccination
Population: as for outcome 3
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
Value | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.59, Parametric correlation; Pearson correlation coefficient = -0.25
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.68, Parametric correlation; Pearson correlation coefficient = -0.12 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.12, Parametric correlation; Pearson correlation coefficient = 0.36
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.26, Parametric correlation; Pearson correlation coefficient = 0.22 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.08, Parametric correlation; Pearson correlation coefficient = 0.43
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.42, Parametric correlation; Pearson correlation coefficient = -0.17 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.02, Parametric correlation; Pearson correlation coefficient = 0.77
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.65, Parametric correlation; Pearson correlation coefficient = -0.12 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.58, Non-parametric correlation; Spearman correlation coefficient = -0.25
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = -0.51, Non-parametric correlation; Spearman correlation coefficient = -0.19 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.24, Non-parametric correlation; Spearman correlation coefficient = 0.28
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.06, Non-parametric correlation; Spearman correlation coefficient = 0.36 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.001, Non-parametric correlation; Spearman correlation coefficient = 0.72
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.12, Non-parametric correlation; Spearman correlation coefficient = -0.32 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.18, Non-parametric correlation; Spearman correlation coefficient = 0.49
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.34, Non-parametric correlation; Spearman correlation coefficient = -0.25 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.06
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; Regression, Linear; R-square = 0.01 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.13
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; Regression, Linear; R-square = 0.05 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.19
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; Regression, Linear; R-square = 0.03 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.60
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 23]; Test type: Superiority or Other; Regression, Linear; R-square = 0.01 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 25: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.001, Parametric correlation; Pearson correlation coefficient = 0.83
Statistical Analysis 26: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p = 0.57, Parametric correlation; Pearson correlation coefficient = 0.14 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 27: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.001, Parametric correlation; Pearson correlation coefficient = 0.65
Statistical Analysis 28: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 27]; Test type: Superiority or Other; p = 0.11, Parametric correlation; Pearson correlation coefficient = 0.31 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 29: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.94, Parametric correlation; Pearson correlation coefficient = -0.02
Statistical Analysis 30: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 1.00, Parametric correlation; Pearson correlation coefficient = -0.0003 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 31: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 1.00, Parametric correlation; Pearson correlation coefficient = 0.004
Statistical Analysis 32: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; p = 0.37, Parametric correlation; Pearson correlation coefficient = -0.30 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 33: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.09, Non-parametric correlation; Spearman correlation coefficient = 0.52
Statistical Analysis 34: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.40, Non-parametric correlation; Spearman correlation coefficient = 0.21 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 35: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.20, Non-parametric correlation; Spearman correlation coefficient = 0.28
Statistical Analysis 36: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 35]; Test type: Superiority or Other; p = 0.03, Non-parametric correlation; Spearman correlation coefficient = 0.41 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 37: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.07, Non-parametric correlation; Spearman correlation coefficient = 0.48
Statistical Analysis 38: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; p = 0.30, Non-parametric correlation; Spearman correlation coefficient = 0.22 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 39: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.74, Non-parametric correlation; Spearman correlation coefficient = 0.26
Statistical Analysis 40: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 39]; Test type: Superiority or Other; p = 0.25, Non-parametric correlation; Spearman correlation coefficient = -0.378 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 41: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.69
Statistical Analysis 42: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 41]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 43: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.42
Statistical Analysis 44: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; Regression, Linear; R-square = 0.10 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 45: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.0004
Statistical Analysis 46: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 45]; Test type: Superiority or Other; Regression, Linear; R-square = 0.00 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 47: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers rise from pre-booster to one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.000
Statistical Analysis 48: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 47]; Test type: Superiority or Other; Regression, Linear; R-square = 0.90 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 49: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.86, Parametric correlation; Pearson correlation coefficient = -0.04
Statistical Analysis 50: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.7, Parametric correlation; Pearson correlation coefficient = 0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 51: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.58, Parametric correlation; Pearson correlation coefficient = -0.11
Statistical Analysis 52: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 51]; Test type: Superiority or Other; p = 0.44, Parametric correlation; Pearson correlation coefficient = -0.13 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 53: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.75, Parametric correlation; Pearson correlation coefficient = -0.07
Statistical Analysis 54: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 53]; Test type: Superiority or Other; p = 0.84, Parametric correlation; Pearson correlation coefficient = -0.04 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 55: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.67, Parametric correlation; Pearson correlation coefficient = -0.11
Statistical Analysis 56: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 55]; Test type: Superiority or Other; p = 0.99, Parametric correlation; Pearson correlation coefficient = -0.002 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 57: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.62, Non-parametric correlation; Spearman correlation coefficient = 0.11
Statistical Analysis 58: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.36, Non-parametric correlation; Spearman correlation coefficient = 0.17 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 59: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.99, Non-parametric correlation; Spearman correlation coefficient = -0.003
Statistical Analysis 60: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 59]; Test type: Superiority or Other; p = 0.24, Non-parametric correlation; Spearman correlation coefficient = -0.20 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 61: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.62, Non-parametric correlation; Spearman correlation coefficient = 0.11
Statistical Analysis 62: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 61]; Test type: Superiority or Other; p = 0.69, Non-parametric correlation; Spearman correlation coefficient = 0.08 — Values from Group 2 and 3 were combined for the analysis
Statistical Analysis 63: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.60, Non-parametric correlation; Spearman correlation coefficient = -0.13
Statistical Analysis 64: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 63]; Test type: Superiority or Other; p = 0.95, Non-parametric correlation; Spearman correlation coefficient = -0.01 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 65: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.0015
Statistical Analysis 66: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 65]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0057 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 67: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 68: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 67]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Groups 2 and 3 were combined for this analysis
Statistical Analysis 69: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.0048
Statistical Analysis 70: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 69]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0018 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 71: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise from pre-booster levels in serogroup specific IgG concentration one month after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 72: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0000 — Values from Group 2 and 3 were combined for this analysis

5. Secondary Outcome: Memory B Cells 1 Month After Primary Vaccination and 1 Week After Third Vaccination by Serogroup A, C, W-135 and Y
Description: Memory B cell response at 1 month after primary vaccination and at 1 week after third vaccination was measured as mean number of meningococcal serogroup specific memory B cells by ELISpot assay per 2x100000 LOC.
  Plasma B cell response at 1 week after vaccination was measured as the mean number of cells secreting antibodies specific for meningococcal serogroup A, C, W-135 and Y, measured by ELISpot assay, per 2x100000 PBMC.
  Serogroup A, C, W-135 and Y specific IgG were measured by ELISA and hSBA GMTs were measured at 1 week after third vaccination.
Time Frame: One month after primary vaccination and 1 week after third vaccination
Population: This outcome was assessed in Group 3 subjects only as they provided a blood draw at 1 week following the MenACWY-CRM booster vaccination. Analysis was performed on PP booster population.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 0 | 0 | 42
Value |  |  | NA — Outcomes are based on correlation and regression coefficients.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.68, Parametric correlation; Pearson correlation coefficient = -0.14
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.09, Parametric correlation; Pearson correlation coefficient = 0.44
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.69, Parametric correlation; Pearson correlation coefficient = 0.11
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.20, Parametric correlation; Pearson correlation coefficient = 0.38
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.88, Non-parametric correlation; Spearman correlation coefficient = -0.05
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.12, Non-parametric correlation; Spearman correlation coefficient = 0.41
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.37, Non-parametric correlation; Spearman correlation coefficient = 0.25
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.36, Non-parametric correlation; Spearman correlation coefficient = 0.28
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.02
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.20
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific plasma cells one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.15
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and memory B cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Parametric correlation; Pearson correlation coefficient = 1.0
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and memory B cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Non-parametric correlation; Spearman correlation coefficient = 1.0
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 1.0
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.0
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and memory B cells one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.0
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.79, Parametric correlation; Pearson correlation coefficient = -0.08
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.16, Parametric correlation; Pearson correlation coefficient = 0.35
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.10, Parametric correlation; Pearson correlation coefficient = 0.48
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.003, Parametric correlation; Pearson correlation coefficient = 0.98
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.91, Non-parametric correlation; Spearman correlation coefficient = -0.03
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.01, Non-parametric correlation; Spearman correlation coefficient = 0.57
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.19, Non-parametric correlation; Spearman correlation coefficient = 0.39
Statistical Analysis 25: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.04, Non-parametric correlation; Spearman correlation coefficient = 0.89
Statistical Analysis 26: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 27: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.12
Statistical Analysis 28: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.23
Statistical Analysis 29: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.96
Statistical Analysis 30: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.46, Parametric correlation; Pearson correlation coefficient = 0.18
Statistical Analysis 31: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.90, Parametric correlation; Pearson correlation coefficient = -0.03
Statistical Analysis 32: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.008, Parametric correlation; Pearson correlation coefficient = 0.51
Statistical Analysis 33: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.08, Parametric correlation; Pearson correlation coefficient = 0.42
Statistical Analysis 34: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup A; Test type: Superiority or Other; p = 0.52, Non-parametric correlation; Spearman correlation coefficient = 0.15
Statistical Analysis 35: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup C; Test type: Superiority or Other; p = 0.18, Non-parametric correlation; Spearman correlation coefficient = 0.27
Statistical Analysis 36: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; p = 0.07, Non-parametric correlation; Spearman correlation coefficient = 0.37
Statistical Analysis 37: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; p = 0.55, Non-parametric correlation; Spearman correlation coefficient = 0.14
Statistical Analysis 38: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.03
Statistical Analysis 39: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.0007
Statistical Analysis 40: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.27
Statistical Analysis 41: Comparison: MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration one week after booster vaccination for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.17

6. Secondary Outcome: CRM197 Specific Memory B Cells 1 Month After Primary Vaccination and at 12 Months of Age and One Month After MenACWY-CRM Third Vaccination
Description: CRM197 specific memory B cell response at each time point was measured as mean number of CRM197 specific memory B cells by ELISpot assay per 2x100000 LOC.
  CRM197 specific IgG concentration was measured by ELISA at 12 months of age and one month after MenACWY-CRM booster vaccination.
Time Frame: 5 months (B cells), 12 months and 13 months (B cells and IgG) of age
Population: Analysis was done on the PP primary population and PP booster population.
Measure: Number
Groups:
- MenACWY-CRM + Routine Vaccines (Group 2): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 12 months), and 1 dose each of MMR and Hib (booster) at 13 months.
  This group had an additional blood draw at the time of enrollment.
- MenACWY-CRM + Routine Vaccines (Group 3): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 12 months), and 1 dose each of MMR and Hib (booster) at 13 months of age.
  This group had an additional blood draw at 6-7 days after third dose of MenACWY-CRM.
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM + Routine Vaccines (Group 2) | MenACWY-CRM + Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
Value | NA — Data were not summarized for each group as correlation and regression deal with relationships among two variables measured on each subject rather than a summary measure (e.g. mean) per vaccine group. | NA — Data were not summarized for each group as correlation and regression deal with relationships among two variables measured on each subject rather than a summary measure (e.g. mean) per vaccine group. | NA — Data were not summarized for each group as correlation and regression deal with relationships among two variables measured on each subject rather than a summary measure (e.g. mean) per vaccine group.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Pearson correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells at 12 months of age; Test type: Superiority or Other; p = 0.0006, Parametric correlation; Pearson correlation coefficient = 0.45 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Spearman correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells at 12 months of age; Test type: Superiority or Other; p = 0.0021, Non-parametric correlation; Spearman correlation coefficient = 0.41 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Linear regression coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells at 12 months of age; Test type: Superiority or Other; Regression, Linear; R-square = 0.21 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells 1 month after booster vaccination; Test type: Superiority or Other; p = 0.53, Parametric correlation; Pearson correlation coefficient = -0.15
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Pearson correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells one month after booster vaccination; Test type: Superiority or Other; p = 0.26, Parametric correlation; Pearson correlation coefficient = 0.21 — Values from Groups 1, 2 and 3 were combined for this analysis
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells one month after booster vaccination; Test type: Superiority or Other; p = 0.84, Non-parametric correlation; Spearman correlation coefficient = -0.05
Statistical Analysis 7: Comparison: MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.26, Non-parametric correlation; Spearman Correlation Coefficient = 0.22 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific memory B cells one month after booster vaccination; Test type: Superiority or Other; Regression, Linear; R-square = 0.02
Statistical Analysis 9: Comparison: MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; Regression, Linear; R-square = 0.05 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Pearson correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration at 12 months of age; Test type: Superiority or Other; p < 0.001, Parametric correlation; Pearson correlation coefficient = 0.33 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Spearman correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration at 12 months of age; Test type: Superiority or Other; p < 0.001, Non-parametric correlation; Spearman correlation coefficient = 0.46 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); Linear regression coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration at 12 months of age; Test type: Superiority or Other; p < 0.001, Regression, Linear; R-square = 0.11 — Values from Group 1, 2 and 3 were combined for this analysis
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Pearson correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration one month after booster vaccination; Test type: Superiority or Other; p = 0.06, Parametric correlation; Pearson correlation coefficient = 0.24
Statistical Analysis 14: Comparison: MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, Parametric correlation; Pearson correlation coefficient = 0.50 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Spearman correlation coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration one month after booster vaccination; Test type: Superiority or Other; p = 0.01, Non-parametric correlation; Spearman correlation coefficient = 0.31
Statistical Analysis 16: Comparison: MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p = 0.10, Non-parametric correlation; Spearman correlation coefficient = 0.20 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between CRM197 specific memory B cells one month after primary vaccination and CRM197 specific IgG concentration one month after booster vaccination; Test type: Superiority or Other; Regression, Linear; R-square = 0.06
Statistical Analysis 18: Comparison: MenACWY-CRM + Routine Vaccines (Group 2) vs MenACWY-CRM + Routine Vaccines (Group 3); [analysis description as in outcome 6, analysis 17]; Test type: Superiority or Other; Regression, Linear; R-square = 0.25 — Values from Group 2 and 3 were combined for this analysis

7. Secondary Outcome: Increase in Serogroup A, C, W-135 and Y Specific Memory B Cells Before and 1 Month After MenACWY-CRM Booster Vaccination at 12 Months of Age Administered Concomitantly With Pneumococcal Conjugate Vaccine or Alone
Description: Memory B cell response before and one month after MenACWY-CRM booster vaccination at 12 months of age was measured as mean number of meningococcal serogroup A, C, W-135 and Y specific memory B cells by ELISpot assay per 2x100000 LOC.
Time Frame: Before and one month after booster vaccination
Population: Analysis was performed on the PP dataset of booster vaccination.
Measure: Mean (Standard Deviation); unit: B cells per 2x100000 lymphocytes
Groups:
- MenACWY-CRM and Routine Vaccines (Group 2): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 13 months), and 1 dose each of MMR and Hib (booster) at 13 months.
  This group had an additional blood draw at the time of enrollment.
- MenACWY-CRM and Routine Vaccines (Group 3): Infants received 2 doses of MenACWY-CRM (at 2 and 4 months) as a primary course of vaccination and third dose (at 12 months) as a booster. Infants also received routine vaccines - 3 doses of DTaP-Hib-IPV (at 2, 3, and 4 months), 3 doses of PCV (at 2, 4, and 13 months), and 1 dose each of MMR and Hib (booster) at 13 months of age.
  This group had an additional blood draw at 6-7 days after third dose of MenACWY-CRM.
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
B cells per 2x100000 lymphocytes
  Serogroup A specific B cells (N=58,29,31) before | 1.811 (1.935) | 1.988 (1.881) | 1.692 (1.398)
  Serogroup A specific B cells (N=54,26,33) after | 6.429 (6.365) | 6.527 (5.957) | 7.488 (12.512)
  Serogroup C specific B cells (N=75,35,38) before | 2.076 (1.926) | 1.983 (1.482) | 2.188 (2.004)
  Serogroup C specific B cells (N=73,37,40) after | 9.437 (10.861) | 8.907 (9.791) | 8.915 (10.830)
  Serogroup W specific B cells (N=75,34,38) before | 1.783 (2.189) | 1.793 (1.531) | 2.067 (2.616)
  Serogroup W specific B cells (N=73,37,39) after | 6.205 (6.776) | 4.430 (5.939) | 5.201 (6.648)
  Serogroup Y specific B cells (N=67,33,34) before | 2.172 (2.934) | 1.556 (0.898) | 1.749 (1.797)
  Serogroup Y specific B cells (N=64,32,34) after | 6.950 (9.122) | 6.603 (8.198) | 5.746 (12.624)

8. Secondary Outcome: Increase in Serogroup A, C, W-135 and Y Specific hSBA Titers Before and 1 Month After MenACWY-CRM Booster Vaccination at 12 Months of Age Administered Concomitantly With Pneumococcal Conjugate Vaccine or Alone
Description: hSBA GMTs were measured before and one month after MenACWY-CRM booster vaccination at 12 months of age.
Time Frame: Before and one month after booster vaccination
Population: Analysis was performed on the PP dataset of booster vaccination.
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
titers
  Serogroup A - hSBA GMT - before | 2.2 [2.05 to 2.36] | 2 [2 to 2] | 2.14 [1.93 to 2.37]
  Serogroup A - hSBA GMT - after | 65 [47 to 89] | 48 [32 to 72] | 67 [44 to 102]
  Serogroup C - hSBA GMT (N=83,39,40)- before | 5.56 [4.23 to 7.3] | 4.83 [3.28 to 7.09] | 5.61 [3.78 to 8.33]
  Serogroup C - hSBA GMT (N=78,39,40)- after | 315 [239 to 417] | 217 [138 to 341] | 308 [214 to 445]
  Serogroup W - hSBA GMT (N=67,37,34)- before | 8.4 [6.03 to 12] | 12 [8.05 to 17] | 10 [6.73 to 15]
  Serogroup W - hSBA GMT (N=67,37,34)- after | 889 [622 to 1271] | 649 [419 to 1004] | 602 [343 to 1057]
  Serogroup Y - hSBA GMT (N=43,25,16)- before | 8.71 [5.82 to 13] | 9.9 [5.39 to 18] | 9.15 [4.95 to 17]
  Serogroup Y - hSBA GMT (N=32,20,15)- after | 492 [305 to 793] | 480 [269 to 857] | 475 [220 to 1025]

9. Secondary Outcome: Serogroups A, C, W-135 and Y Specific Memory B Cell Response in Children Lacking a hSBA Titer of ≥1:8 One Month After MenACWY-CRM Primary Vaccination
Description: The memory B cell response in children lacking a hSBA titer ≥1:8 one month after MenACWY-CRM primary vaccination was calculated as the mean number of meningococcal serogroup specific memory B cells, measured by ELISpot assay per 2x100000 LOC.
Time Frame: One month after primary vaccination
Population: Analysis was performed on the PP primary population and PP persistence population, subjects lacking hSBA ≥1:8 one month after primary vaccination.
Measure: Mean (Standard Deviation); unit: B cells per 2x100000 lymphocytes
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 88 | 34 | 50
B cells per 2x100000 lymphocytes
  Serogroup A specific memory B cells (N=24,11,8) | 1.533 (1.028) | 1.391 (0.467) | 1.250 (0.000)
  Serogroup C specific memory B cells (N=6,2,1) | 2.667 (2.444) | 1.250 (0.000) | 1.250 (NA) — Analysis was done on one subject only
  Serogroup W-135 specific memory B cells (N=3,0,1) | 1.250 (0.000) | NA (NA) — None of the subject had hSBA titer <1:8 | 1.250 (NA) — Analysis was done on one subject only
  Serogroup Y specific memory B cells (N=0,1,1) | NA (NA) — None of the subject had hSBA titer <1:8 | 1.250 (0.000) | 1.250 (0.000)

10. Secondary Outcome: Serogroup A, C, W-135 and Y Specific Memory B Cells and Plasma B Cells After MenACWY-CRM Primary Vaccination
Description: To assess the kinetics of serogroup A, C, W-135 and Y specific memory B cells, plasma B cells and IgG concentrations were measured on days 0, 7, 14, 49, 90, and 120 following vaccination with MenACWY-CRM vaccination at month 4 of the study.
  The memory B cell response at different timepoint was defined as the mean number of meningococcal serogroup A, C, W-135 and Y specific memory B cells, measured in vitro by ELISpot assay per 2x100000 lymphocytes obtained from culture (LOC) of peripheral blood mononuclear cells (PBMC) circulating in blood incubated for 5.5 days in the presence of polyclonal B cell activators in vitro.
  The B plasma cell response at each time point was defined as the mean number of cells secreting antibodies specific for meningococcal serogroup A, C, W-135 and Y, measured by ELISpot assay, per 2x100000 PBMC.
Time Frame: Day 0, 7, 14, 49, 90, and 120 after MenACWY-CRM vaccination at month 4
Population: This outcome was assessed in Group 1 PP set population.
Measure: Mean (Standard Deviation); unit: per 2x100000 cells
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1)
Number analyzed (Participants) | 88
per 2x100000 cells
  Serogroup A sp. memory B cell (N=4)- Day 0 | 1.25 (0)
  Serogroup A sp. memory B cell (N=14)- Day 7 | 3.889 (5.07)
  Serogroup A sp. memory B cell (N=7)- Day 14 | 2.343 (2.891)
  Serogroup A sp. memory B cell (N=10)- Day 49 | 1.97 (1.533)
  Serogroup A sp. memory B cell (N=9)- Day 90 | 1.25 (0)
  Serogroup A sp. memory B cell (N=11)- Day 120 | 1.845 (1.14)
  Serogroup C sp. memory B cell (N=6)- Day 0 | 1.558 (0.775)
  Serogroup C sp. memory B cell (N=16)- Day 7 | 2.856 (2.974)
  Serogroup C sp. memory B cell (N=12)- Day 14 | 5.183 (5.723)
  Serogroup C sp. memory B cell (N=13)- Day 49 | 2.323 (2.044)
  Serogroup C sp. memory B cell (N=16)- Day 90 | 2.469 (1.865)
  Serogroup C sp. memory B cell (N=14)- Day 120 | 1.561 (1.163)
  Serogroup W-135 sp. memory B cell (N=4)- Day 0 | 1.25 (0)
  Serogroup W-135 sp. memory B cell (N=15)- Day 7 | 3.737 (6.68)
  Serogroup W-135 sp. memory B cell (N=12)- Day 14 | 2.754 (2.245)
  Serogroup W-135 sp. memory B cell (N=13)- Day 49 | 2.735 (2.4)
  Serogroup W-135 sp. memory B cell (N=14)- Day 90 | 1.404 (0.575)
  Serogroup W-135 sp. memory B cell (N=14)- Day 120 | 1.25 (0)
  Serogroup Y sp. memory B cell (N=3)- Day 0 | 1.25 (0)
  Serogroup Y sp. memory B cell (N=15)- Day 7 | 4.847 (9.043)
  Serogroup Y sp. memory B cell (N=7)- Day 14 | 1.471 (0.586)
  Serogroup Y sp. memory B cell (N=11)- Day 49 | 1.482 (0.769)
  Serogroup Y sp. memory B cell (N=12)- Day 90 | 1.567 (0.74)
  Serogroup Y sp. memory B cell (N=13)- Day 120 | 1.527 (0.684)
  Serogroup A sp. plasma B cell (N=3)- Day 0 | 1.25 (0)
  Serogroup A sp. plasma B cell (N=1)- Day 7 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup A sp. plasma B cell (N=1)- Day 14 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup A sp. plasma B cell (N=2)- Day 49 | 1.25 (0)
  Serogroup A sp. plasma B cell (N=2)- Day 90 | 1.25 (0)
  Serogroup A sp. plasma B cell (N=2)- Day 120 | 1.25 (0)
  Serogroup C sp. plasma B cell (N=3)- Day 0 | 1.25 (0)
  Serogroup C sp. plasma B cell (N=2)- Day 7 | 2.025 (1.096)
  Serogroup C sp. plasma B cell (N=1)- Day 14 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup C sp. plasma B cell (N=2)- Day 49 | 1.25 (0)
  Serogroup C sp. plasma B cell (N=2)- Day 90 | 1.25 (0)
  Serogroup C sp. plasma B cell (N=3)- Day 120 | 1.25 (0)
  Serogroup W-135 sp. plasma B cell (N=3)- Day 0 | 1.25 (0)
  Serogroup W-135 sp. plasma B cell (N=1)- Day 7 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup W-135 sp. plasma B cell (N=1)- Day 14 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup W-135 sp. plasma B cell (N=2)- Day 49 | 1.25 (0)
  Serogroup W-135 sp. plasma B cell (N=2)- Day 90 | 1.25 (0)
  Serogroup W-135 sp. plasma B cell (N=3)- Day 120 | 1.25 (0)
  Serogroup Y sp. plasma B cell (N=3)- Day 0 | 1.25 (0)
  Serogroup Y sp. plasma B cell (N=1)- Day 7 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup Y sp. plasma B cell (N=1)- Day 14 | 1.25 (NA) — Only one subject was analyzed.
  Serogroup Y sp. plasma B cell (N=2)- Day 49 | 1.25 (0)
  Serogroup Y sp. plasma B cell (N=2)- Day 90 | 1.25 (0)
  Serogroup Y sp. plasma B cell (N=2)- Day 120 | 1.25 (0)

11. Secondary Outcome: Serogroup A, C, W-135 and Y Specific hSBA Titers After MenACWY-CRM Primary Vaccination
Description: To assess the kinetics of serogroup A, C, W-135 and Y specific hSBA titers, the geometric mean titer was measured on day 0, 7, 14, 30, 49, 90, and 120 following vaccination with MenACWY-CRM vaccination at month 4 of the study.
Time Frame: Day 0, 7, 14, 30, 49, 90,120 after MenACWY-CRM vaccination at month 4
Population: This outcome was assessed in Group 1 PP set population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1)
Number analyzed (Participants) | 88
titers
  Serogroup A - hSBA GMTs (N=7)- Day 0 | 2 [2 to 2]
  Serogroup A - hSBA GMTs (N=18)- Day 7 | 13 [7.15 to 25]
  Serogroup A - hSBA GMTs (N=16)- Day 14 | 26 [10 to 63]
  Serogroup A - hSBA GMTs - Day 30 | 9.79 [7.22 to 13]
  Serogroup A - hSBA GMTs (N=16)- Day 49 | 9.53 [4.49 to 20]
  Serogroup A - hSBA GMTs (N=18)- Day 90 | 2.63 [1.77 to 3.91]
  Serogroup A - hSBA GMTs (N=16)- Day 120 | 4.45 [2.25 to 8.83]
  Serogroup C - hSBA GMTs (N=5)- Day 0 | 7.19 [1.33 to 39]
  Serogroup C - hSBA GMTs (N=16)- Day 7 | 138 [43 to 439]
  Serogroup C - hSBA GMTs (N=12)- Day 14 | 180 [55 to 596]
  Serogroup C - hSBA GMTs (N=31)- Day 30 | 105 [73 to 151]
  Serogroup C - hSBA GMTs (N=16)- Day 49 | 104 [50 to 219]
  Serogroup C - hSBA GMTs (N=18)- Day 90 | 31 [18 to 53]
  Serogroup C - hSBA GMTs (N=16)- Day 120 | 15 [6.5 to 36]
  Serogroup W-135 - hSBA GMTs (N=5)- Day 0 | 4.43 [1.48 to 13]
  Serogroup W-135 - hSBA GMTs (N=12)- Day 7 | 99 [42 to 232]
  Serogroup W-135 - hSBA GMTs (N=9)- Day 14 | 144 [42 to 497]
  Serogroup W-135 - hSBA GMTs (N=61)- Day 30 | 60 [44 to 83]
  Serogroup W-135 - hSBA GMTs (N=11)- Day 49 | 35 [18 to 69]
  Serogroup W-135 - hSBA GMTs (N=15)- Day 90 | 20 [11 to 35]
  Serogroup W-135 - hSBA GMTs (N=4)- Day 120 | 12 [7.58 to 20]
  Serogroup Y - hSBA GMTs (N=1)- Day 0 | 2 [NA to NA] — Only one subject was analyzed.
  Serogroup Y - hSBA GMTs (N=8)- Day 7 | 32 [8.06 to 123]
  Serogroup Y - hSBA GMTs (N=4)- Day 14 | 95 [8 to 1131]
  Serogroup Y - hSBA GMTs (N=20)- Day 30 | 24 [16 to 38]
  Serogroup Y - hSBA GMTs (N=8)- Day 49 | 33 [11 to 101]
  Serogroup Y - hSBA GMTs (N=9)- Day 90 | 12 [4.62 to 29]
  Serogroup Y - hSBA GMTs (N=8)- Day 120 | 8.15 [3.77 to 18]

12. Secondary Outcome: Correlation and Linear Regression Coefficients Between Serogroup A, C, W-135 and Y Specific Memory B Cells 1 Month After MenACWY-CRM Primary Vaccination and IgG Concentration at Day 1 in the Serum of Mothers of Infants
Description: The serogroup A, C, W-135 and Y specific IgG concentrations were measured in the serum of mothers at the time of their enrollment into the study (Day 1) by ELISA.
Time Frame: Day 1 (IgG) and one month after primary vaccination (B cells)
Population: Analysis was performed on the PP primary population.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 88 | 34 | 50
Value | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients. | NA — Outcomes are based on correlation and regression coefficients.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup A; Test type: Superiority or Other; p = 0.70, Parametric correlation; Pearson correlation coefficient = 0.04
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup C; Test type: Superiority or Other; p = 0.63, Parametric correlation; Pearson correlation coefficient = -0.04
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup W-135; Test type: Superiority or Other; p = 0.74, Parametric correlation; Pearson correlation coefficient = -0.03
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Pearson correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup Y; Test type: Superiority or Other; p = 0.74, Parametric correlation; Pearson correlation coefficient = -0.03
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup A; Test type: Superiority or Other; p = 0.05, Non-parametric correlation; Spearman correlation coefficient = 0.18
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup C; Test type: Superiority or Other; p = 0.36, Non-parametric correlation; Spearman correlation coefficient = -0.07
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup W-135; Test type: Superiority or Other; p = 0.18, Non-parametric correlation; Spearman correlation coefficient = -0.11
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Spearman correlation coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup Y; Test type: Superiority or Other; p = 0.82, Non-parametric correlation; Spearman correlation coefficient = 0.02
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.0013
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.0014
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.0008
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 1) vs MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at day 1 in the serum of mother for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.0009

13. Secondary Outcome: Linear Regression Coefficients (1) Between Serogroup A, C, W-135 and Y Memory B at 5 Months and hSBA Titers at 12 Months, (2) Between Serogroup A, C, W-135 and Y Memory B at 5 Months and IgG at 12 Months, After a 2-Dose Primary Course of MenACWY-CRM
Description: Linear regression analysis between memory B cells at 5 months of age and hSBA titers and IgG at 12 months of age was performed with and without inclusion of demographic factors (subject's household smoking status, number of older children living in subject's household, attendance at daycare and total duration of breast feeding) in the model.
Time Frame: 1 month post primary vaccination (B cells) and 12 months (hSBA titers and IgG)
Population: Analysis was performed on the PP dataset of persistence population.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 79 | 37 | 39
Value | NA — Outcomes are based on regression coefficient. | NA — Outcomes are based on regression coefficient. | NA — Outcomes are based on regression coefficient.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.34
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; Regression, Linear; R-square = 0.14 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells at 5 months of age and hSBA titers at 12 months of age after a 2, 4-month course of MenACWY-CRM vaccination for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.09
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.16 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.22
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 5]; Test type: Superiority or Other; Regression, Linear; R-square = 0.33 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.74
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; Regression, Linear; R-square = 0.53 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.37
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 9]; Test type: Superiority or Other; Regression, Linear; R-square = 0.14 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.13
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 11]; Test type: Superiority or Other; Regression, Linear; R-square = 0.17 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.9
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; Regression, Linear; R-square = 0.78 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and hSBA titers at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.94
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 15]; Test type: Superiority or Other; Regression, Linear; R-square = 0.85 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.03
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 17]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.0070
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; Regression, Linear; R-square = 0.04 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.02
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 21]; Test type: Superiority or Other; Regression, Linear; R-square = 0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.13
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 23]; Test type: Superiority or Other; Regression, Linear; R-square = 0.28 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 25: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.3
Statistical Analysis 26: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; Regression, Linear; R-square = 0.1 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 27: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.11
Statistical Analysis 28: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 27]; Test type: Superiority or Other; Regression, Linear; R-square = 0.06 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 29: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.17
Statistical Analysis 30: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 29]; Test type: Superiority or Other; Regression, Linear; R-square = 0.21 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 31: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors memory B cells one month after primary vaccination and serogroup specific IgG concentration at 12 months of age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.39
Statistical Analysis 32: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 13, analysis 31]; Test type: Superiority or Other; Regression, Linear; R-square = 0.33 — Values from Group 2 and 3 were combined for this analysis

14. Secondary Outcome: Linear Regression Coefficients (1) Between Serogroup A, C, W-135 and Y Memory B Cells at 5 Months and Rise in hSBA Titers, (2) Between Serogroup A, C, W-135 and Y Memory B Cells at 5 Months and Rise in IgG, After Third Dose of MenACWY-CRM at 12 Months
Description: The rise in serogroup-specific hSBA and IgG was calculated by pre/post third dose geometric mean ratios, calculated by the difference in the log10 of the concentrations/titers measured at 13 months to the log10 of the concentrations at 12 months: i.e. rise = log10(x) at 13 months minus log10(x) at 12 months where x is the serogroup specific IgG or SBA titers.
  Linear regression analysis between memory B cells at 5 months of age and rise in hSBA titers or IgG at 12 months of age was performed with and without inclusion of demographic factors (subject's household smoking status, number of older children living in subject's household, attendance at daycare and total duration of breast feeding) in the model.
Time Frame: 1 month post primary vaccination (B cells) and 12 months (hSBA titers and IgG)
Population: Analysis was performed on the PP dataset after booster vaccination.
Measure: Number
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
Value | NA — Outcomes are based on linear regression coefficient. | NA — Outcomes are based on linear regression coefficient. | NA — Outcomes are based on linear regression coefficient.
Statistical Analysis 1: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.24
Statistical Analysis 2: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Regression, Linear; R-square = 0.19 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 3: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.52
Statistical Analysis 4: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; Regression, Linear; R-square = 0.07 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 5: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 1
Statistical Analysis 6: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 5]; Test type: Superiority or Other; Regression, Linear; R-square = 0.29 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 7: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.19
Statistical Analysis 8: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; Regression, Linear; R-square = 0.05 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 9: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.7
Statistical Analysis 10: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 9]; Test type: Superiority or Other; Regression, Linear; R-square = 0.21 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 11: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.5
Statistical Analysis 12: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 11]; Test type: Superiority or Other; Regression, Linear; R-square = 0.16 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 13: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 1
Statistical Analysis 14: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; Regression, Linear; R-square = 0.3 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 15: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in hSBA after booster vaccination age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.21
Statistical Analysis 16: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 15]; Test type: Superiority or Other; Regression, Linear; R-square = 0.12 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 17: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.0015
Statistical Analysis 18: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 17]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0057 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 19: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 20: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; Regression, Linear; R-square = 0.02 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 21: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup W-135; Test type: Superiority or Other; Regression, Linear; R-square = 0.0048
Statistical Analysis 22: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 21]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0018 — Values from Groups 2 and 3 were combined for this analysis
Statistical Analysis 23: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.01
Statistical Analysis 24: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; Regression, Linear; R-square = 0.0000 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 25: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup A; Test type: Superiority or Other; Regression, Linear; R-square = 0.27
Statistical Analysis 26: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; Regression, Linear; R-square = 0.19 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 27: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup C; Test type: Superiority or Other; Regression, Linear; R-square = 0.08
Statistical Analysis 28: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 27]; Test type: Superiority or Other; Regression, Linear; R-square = 0.08 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 29: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup W-135; Test type: Superiority or Other; p = 0.0436, Regression, Linear; R-square = 0.45
Statistical Analysis 30: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 29]; Test type: Superiority or Other; Regression, Linear; R-square = 0.17 — Values from Group 2 and 3 were combined for this analysis
Statistical Analysis 31: Comparison: MenACWY-CRM and Routine Vaccines (Group 1); Linear regression coefficient between demographic factors, memory B cells one month after primary vaccination and rise in serogroup specific IgG concentration after booster vaccination age for the serogroup Y; Test type: Superiority or Other; Regression, Linear; R-square = 0.37
Statistical Analysis 32: Comparison: MenACWY-CRM and Routine Vaccines (Group 2) vs MenACWY-CRM and Routine Vaccines (Group 3); [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; Regression, Linear; R-square = 0.07 — Values from Group 2 and 3 were combined for this analysis

15. Secondary Outcome: Percentage of Subjects Who Reported Injection Site Local Reactions After Each MenACWY-CRM and Routine Infant Vaccinations.
Description: Safety was assessed as the percentage of subjects who reported injection site local reactions during 7-day follow-up period after each MenACWY-CRM and routine infant vaccination administered as a primary course of vaccination.
Time Frame: 7 days post each MenACWY-CRM and routine infant vaccination
Population: The analysis was performed on the Safety Population.
Measure: Number; unit: Percentage of subjects
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 108 | 54 | 54
Percentage of subjects
  Tenderness - MenACWY-CRM (Vaccination 1) | 32 | 35 | 22
  Tenderness - MenACWY-CRM (Vaccination 2) | 19 | 28 | 17
  Erythema - MenACWY-CRM (Vaccination 1) | 94 | 96 | 94
  Erythema - MenACWY-CRM (Vaccination 2) | 96 | 96 | 100
  Induration - MenACWY-CRM (Vaccination 1) | 35 | 37 | 39
  Induration - MenACWY-CRM (Vaccination 2) | 44 | 50 | 54
  Tenderness - DTaP-IPV-Hib (Vaccination 1) | 40 | 43 | 28
  Tenderness - DTaP-IPV-Hib (Vaccination 2) | 31 | 35 | 31
  Tenderness - DTaP-IPV-Hib (Vaccination 3) | 27 | 33 | 24
  Erythema - DTaP-IPV-Hib (Vaccination 1) | 97 | 98 | 91
  Erythema - DTaP-IPV-Hib (Vaccination 2) | 94 | 93 | 100
  Erythema - DTaP-IPV-Hib (Vaccination 3) | 97 | 98 | 98
  Induration - DTaP-IPV-Hib (Vaccination 1) | 49 | 50 | 54
  Induration - DTaP-IPV-Hib (Vaccination 2) | 53 | 65 | 54
  Induration - DTaP-IPV-Hib (Vaccination 3) | 66 | 72 | 70
  Tenderness - PCV (Vaccination 1) | 40 | 39 | 33
  Tenderness - PCV (Vaccination 2) | 27 | 39 | 26
  Erythema - PCV (Vaccination 1) | 95 | 98 | 93
  Erythema - PCV (Vaccination 2) | 97 | 96 | 100
  Induration - PCV (Vaccination 1) | 38 | 44 | 50
  Induration - PCV (Vaccination 2) | 53 | 61 | 65

16. Secondary Outcome: Percentage of Subjects Who Reported Solicited Systemic Reactions After MenACWY-CRM and Routine Infants Primary Vaccinations
Description: Safety was assessed as the percentage of subjects who reported systemic reactions during 7-day follow-up period after MenACWY-CRM (2 and 4 months) and routine infant primary vaccinations (2, 3 and 4 months).
Time Frame: 7 days post vaccination at 2, 3, and 4 months of age
Population: The analysis was performed on the safety population.
Measure: Number; unit: Percentage of subjects
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 108 | 54 | 54
Percentage of subjects
  Change in eat. habits (N=106,54,54)- Vaccination 1 | 19 | 20 | 30
  Change in eat. habits (N=107,53,54)- Vaccination 2 | 18 | 15 | 17
  Change in eat. habits (N=106,54,53)- Vaccination 3 | 19 | 26 | 30
  Sleepiness (Vaccination 1) | 58 | 54 | 59
  Sleepiness (Vaccination 2) | 39 | 33 | 52
  Sleepiness (Vaccination 3) | 35 | 33 | 37
  Vomiting (Vaccination 1) | 24 | 11 | 17
  Vomiting (Vaccination 2) | 14 | 13 | 6
  Vomiting (Vaccination 3) | 15 | 11 | 15
  Diarrhea (Vaccination 1) | 20 | 20 | 15
  Diarrhea (Vaccination 2) | 17 | 9 | 13
  Diarrhea (Vaccination 3) | 9 | 17 | 13
  Irritability (Vaccination 1) | 66 | 69 | 61
  Irritability (Vaccination 2) | 47 | 76 | 50
  Irritability (Vaccination 3) | 51 | 56 | 57
  Unusual crying (Vaccination 1) | 27 | 20 | 15
  Unusual crying (Vaccination 2) | 17 | 28 | 19
  Unusual crying (Vaccination 3) | 21 | 15 | 26
  Fever (≥38 °C) - Vaccination 1 | 4 | 4 | 0
  Fever (≥38 °C) - Vaccination 2 | 6 | 6 | 0
  Fever (≥38 °C) - Vaccination 3 | 6 | 9 | 4
  Analg. Antipyr. Med. Used (Vaccination 1) | 40 | 26 | 28
  Analg. Antipyr. Med. Used (Vaccination 2) | 26 | 44 | 39
  Analg. Antipyr. Med. Used (Vaccination 3) | 41 | 33 | 56

17. Secondary Outcome: Percentage of Subjects Who Reported Injection Site Local Reactions After MenACWY-CRM and PCV Vaccinations at 12 Months of Age
Description: Safety was assessed as the percentage of subjects who reported injection site local reactions during 7-day follow-up period after MenACWY-CRM and PCV vaccinations at 12 months of age.
Time Frame: 7 days post 12 month vaccination
Population: The analysis was performed on safety after booster population (safety population who received vaccination at 12 months of age).
Measure: Number; unit: Percentage of subjects
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 103 | 50 | 52
Percentage of subjects
  Tenderness - MenACWY-CRM | 28 | 28 | 19
  Erythema - MenACWY-CRM | 99 | 92 | 94
  Induration - MenACWY-CRM | 52 | 50 | 56
  Tenderness - PCV | 0 | 30 | 21
  Erythema - PCV | 0 | 86 | 94
  Induration - PCV | 0 | 48 | 63

18. Secondary Outcome: Percentage of Subjects Who Reported Solicited Systemic Reactions After MenACWY-CRM and PCV Vaccination at 12 Months of Age
Description: Safety was assessed as the percentage of subjects who reported systemic reactions during 7-day follow-up period after MenACWY-CRM and PCV vaccination at 12 months of age.
Time Frame: 7 days post 12 months vaccination
Population: as for outcome 17
Measure: Number; unit: Percentage of subjects
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 103 | 50 | 52
Percentage of subjects
  Change in eating habits (N=97,48,52) | 23 | 23 | 31
  Sleepiness | 20 | 24 | 25
  Vomiting | 3 | 10 | 12
  Diarrhea | 14 | 16 | 15
  Irritability | 25 | 46 | 40
  Unusual crying | 12 | 20 | 15
  Fever (≥38 °C) | 8 | 6 | 6
  Analgesics Antipyretics Medicine Used | 32 | 44 | 46

19. Secondary Outcome: Increase in Serogroup A, C, W-135 and Y Specific IgG Concentrations Before and 1 Month After MenACWY-CRM Booster Vaccination at 12 Months of Age Administered Concomitantly With Pneumococcal Conjugate Vaccine or Alone
Description: Serogroup A, C, W-135 and Y specific IgG concentrations were measured before and one month after MenACWY-CRM booster vaccination by ELISA.
Time Frame: Before and one month after booster vaccination
Population: Analysis was performed on the PP dataset of booster vaccination.
Measure: Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Number analyzed (Participants) | 85 | 40 | 42
µg/mL
  Serogroup A specific IgG (N=49,23,47) before | 0.37 [0.27 to 0.49] | 0.33 [0.23 to 0.46] | 0.31 [0.23 to 0.42]
  Serogroup A specific IgG (N=66,34,38) after | 4.59 [3.63 to 5.89] | 3.5 [2.6 to 4.73] | 5.18 [3.84 to 6.99]
  Serogroup C specific IgG (N=55,25,26) before | 0.19 [0.16 to 0.23] | 0.18 [0.14 to 0.22] | 0.2 [0.15 to 0.28]
  Serogroup C specific IgG (N=59,33,37) after | 1.83 [1.43 to 2.35] | 1.67 [1.18 to 2.36] | 2.63 [1.87 to 3.7]
  Serogroup W specific IgG (N=55,21,26) before | 0.31 [0.25 to 0.38] | 0.35 [0.25 to 0.48] | 0.29 [0.2 to 0.43]
  Serogroup W specific IgG (N=56,32,32) after | 5.97 [4.67 to 7.64] | 5.37 [4.06 to 7.1] | 5.12 [3.5 to 7.5]
  Serogroup Y specific IgG (N=49,21,24) before | 0.43 [0.34 to 0.55] | 0.47 [0.33 to 0.67] | 0.37 [0.25 to 0.55]
  Serogroup Y specific IgG (N=56,31,33) after | 6.2 [4.77 to 8.05] | 5.58 [4.06 to 7.67] | 5.75 [3.93 to 8.42]

20. Secondary Outcome: Serogroup A, C, W-135 and Y Specific IgG Concentrations After MenACWY-CRM Primary Vaccination
Description: To assess the kinetics of serogroup A, C, W-135 and Y specific IgG concentrations, the geometric mean concentration was measured on day 0, 7, 14, 30, 49, 90, and 120 following vaccination with MenACWY-CRM vaccination at month 4 of the study.
Time Frame: Day 0, 7, 14, 30, 49, 90,120 after MenACWY-CRM vaccination at month 4
Population: This outcome was assessed in Group 1 PP set population.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1)
Number analyzed (Participants) | 88
µg/mL
  Serogroup A specific IgG (N=3)- Day 0 | 0.98 [0.0094 to 1.01]
  Serogroup A specific IgG (N=9)- Day 7 | 2.23 [1.02 to 4.87]
  Serogroup A specific IgG (N=7)- Day 14 | 2.27 [0.75 to 6.9]
  Serogroup A specific IgG (N=45)- Day 30 | 1.29 [1.01 to 1.65]
  Serogroup A specific IgG (N=5)- Day 49 | 1.39 [0.47 to 4.14]
  Serogroup A specific IgG (N=5)- Day 90 | 0.94 [0.62 to 1.43]
  Serogroup A specific IgG (N=1)- Day 120 | 1.03 [NA to NA] — only one subject was analyzed
  Serogroup C specific IgG (N=4)- Day 0 | 0.92 [0.19 to 4.35]
  Serogroup C specific IgG (N=14)- Day 7 | 1.4 [0.85 to 2.28]
  Serogroup C specific IgG (N=8)- Day 14 | 1.43 [0.76 to 2.7]
  Serogroup C specific IgG (N=60)- Day 30 | 0.94 [0.77 to 1.14]
  Serogroup C specific IgG (N=5)- Day 49 | 1.02 [0.28 to 3.69]
  Serogroup C specific IgG (N=7)- Day 90 | 0.75 [0.46 to 1.23]
  Serogroup C specific IgG (N=5)- Day 120 | 0.85 [0.26 to 2.75]
  Serogroup W-135 specific IgG (N=3)- Day 0 | 0.43 [0.0096 to 1.9]
  Serogroup W-135 specific IgG (N=10)- Day 7 | 3.75 [1.76 to 8]
  Serogroup W-135 specific IgG (N=8)- Day 14 | 3.77 [1.82 to 7.84]
  Serogroup W-135 specific IgG (N=39)- Day 30 | 1.53 [1.14 to 2.05]
  Serogroup W-135 specific IgG (N=6)- Day 49 | 2.58 [0.83 to 8.05]
  Serogroup W-135 specific IgG (N=9)- Day 90 | 0.81 [0.59 to 1.13]
  Serogroup W-135 specific IgG (N=2)- Day 120 | 0.57 [0.0011 to 3.05]
  Serogroup Y specific IgG (N=3)- Day 0 | 0.82 [0.039 to 18]
  Serogroup Y specific IgG (N=4)- Day 7 | 1.46 [0.24 to 8.99]
  Serogroup Y specific IgG (N=3)- Day 14 | 5.04 [0.58 to 44]
  Serogroup Y specific IgG (N=33)- Day 30 | 1.34 [1.01 to 1.79]
  Serogroup Y specific IgG (N=3)- Day 49 | 2.47 [0.24 to 26]
  Serogroup Y specific IgG (N=2)- Day 90 | 0.57 [0.039 to 8.17]

ADVERSE EVENTS:
Time Frame: All the serious adverse events were collected throughout the study (day 1 to 18 months).
Description: Other adverse events included solicited local and systemic reactions and non-serious unsolicited adverse events.
  Solicited local and systemic reactions were collected from day 1 to day 7 after each vaccination.
  Non-serious unsolicited adverse events were collected from 7 days after each vaccination to the next visit.
Arm/Group | MenACWY-CRM and Routine Vaccines (Group 1) | MenACWY-CRM and Routine Vaccines (Group 2) | MenACWY-CRM and Routine Vaccines (Group 3)
Serious Adverse Events (participants affected / at risk) | 7/108 | 4/54 | 6/54
Other Adverse Events (participants affected / at risk) | 108/108 | 54/54 | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM and Routine Vaccines (Group 1) (N=108) | MenACWY-CRM and Routine Vaccines (Group 2) (N=54) | MenACWY-CRM and Routine Vaccines (Group 3) (N=54)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM and Routine Vaccines (Group 1) (N=108) | MenACWY-CRM and Routine Vaccines (Group 2) (N=54) | MenACWY-CRM and Routine Vaccines (Group 3) (N=54)
Conjunctivitis (Eye disorders) | 7 (7) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 45 (45) | 23 (23) | 19 (19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2)
Teething (Gastrointestinal disorders) | 14 (14) | 8 (8) | 5 (5)
Vomiting (Gastrointestinal disorders) | 43 (43) | 20 (20) | 19 (19)
Erythema (General disorders) | 108 (108) | 53 (53) | 54 (54)
Induration (General disorders) | 91 (91) | 50 (50) | 50 (50)
Pain (General disorders) | 74 (74) | 42 (42) | 38 (38)
Irritability (General disorders) | 93 (93) | 53 (53) | 47 (47)
Pyrexia (General disorders) | 25 (25) | 12 (12) | 9 (9)
Ear infection (Infections and infestations) | 7 (7) | 5 (5) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 10 (10) | 11 (11) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 21 (21) | 15 (15) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2) | 6 (6)
Crying (Nervous system disorders) | 49 (49) | 29 (29) | 29 (29)
Somnolence (Nervous system disorders) | 81 (81) | 40 (40) | 42 (42)
Eating disorder (Psychiatric disorders) | 55 (55) | 30 (30) | 31 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 6 (6) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
the terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.